CLINICAL TRIAL: NCT01674374
Title: A Phase 2 Placebo Controlled Randomized Study of the Effect of SAMITAL on Severity and Duration of Mucositis Induced by Chemoradiation for Head and Neck Cancer (HNC)
Brief Title: Botanical Therapy in Treating Mucositis in Patients With Head and Neck Cancer Who Have Undergone Chemoradiation Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: I 184910; NCI-2012-01030 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-08-02; First posted 2012-08-28 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Mucositis; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Mucositis; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Vaccinium myrtillus extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (SAMITAL) (Experimental): Beginning as soon as symptoms arise during chemoradiotherapy, patients receive Vaccinium myrtillus extract/Macleaya cordata alkaloids/Echinacea angustifolia extract granules PO QID. Patients may continue to receive Vaccinium myrtillus extract/Macleaya cordata alkaloids/Echinacea angustifolia extract granules for up to 4 weeks after completion of radiation therapy for a maximum of 11 weeks.
  Interventions: Procedure: quality-of-life assessment; Other: questionnaire administration; Drug: Vaccinium myrtillus/Macleaya cordata/Echinacea angustifolia extract granules
- Arm II (placebo) (Placebo Comparator): Beginning as soon as symptoms arise during chemoradiotherapy, patients receive placebo PO QID. Patients may continue to receive placebo for up to 4 weeks after completion of radiation therapy for a maximum of 11 weeks.
  Interventions: Other: placebo; Procedure: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies
Drug: Vaccinium myrtillus/Macleaya cordata/Echinacea angustifolia extract granules — Given PO
  Other Names: Samital granules; V. myrtillus/M. cordata/E. angustfolia granules
  Arms: Arm I (SAMITAL)

SUMMARY:
The purpose of this study is to find out what effects (good and bad) SAMITAL (Vaccinium myrtillus extract/Macleaya cordata alkaloids/Echinacea angustifolia extract granules) has on the management of mucositis (inflammation and ulceration that occurs in the mouth) brought on by chemotherapy and radiation therapy for squamous cell carcinoma of the head and neck

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the tolerability of SAMITAL granules for suspension. II. To assess the efficacy of SAMITAL granules for suspension in reducing the incidence of severe mucositis (World Health Organization [WHO] mucositis scale score of 3 or 4) induced by concurrent chemoradiation for head and neck cancer (HNC).

SECONDARY OBJECTIVES:

I. To assess the effect of SAMITAL granules for suspension on the severity and duration of mucositis (WHO mucositis scale and patient self-assessment with the Oral Mucositis Daily Questionnaire [OMDQ]).

II. To assess the effect of SAMITAL granules for suspension on validated patient reported quality of life measures (European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire [QLQ]-C30 and EORTC QLQ Head and Neck Cancer Specific Module).

III. To assess the rate of any grade 3 - grade 4 infections. IV. To assess the cumulative dose of opioids needed. V. To assess weight loss and need for tube feeding. VI. To assess treatment breaks and/or chemotherapy dose reduction.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Beginning as soon as symptoms arise during chemoradiotherapy, patients receive Vaccinium myrtillus extract/Macleaya cordata alkaloids/Echinacea angustifolia extract granules orally (PO) four times daily (QID). Patients may continue to receive Vaccinium myrtillus extract/Macleaya cordata alkaloids/Echinacea angustifolia extract granules for up to 4 weeks after completion of radiation therapy for a maximum of 11 weeks.

ARM II: Beginning as soon as symptoms arise during chemoradiotherapy, patients receive placebo PO QID. Patients may continue to receive placebo for up to 4 weeks after completion of radiation therapy for a maximum of 11 weeks.

After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients with no distant metastatic disease
* Have histologically proven diagnosis of squamous cell carcinoma (stage III - IV) of the paranasal sinuses, nasopharynx, larynx, hypopharynx, oral cavity and/or oropharynx; treated with definitive concurrent chemoradiotherapy; OR histologically proven diagnosis of squamous cell carcinoma of the paranasal sinuses, nasopharynx, larynx, hypopharynx, or oropharynx with finding of need for concurrent chemoradiotherapy (extracapsular extension, positive surgical margin, more than one lymph node positive, stage III - IV disease, perineural invasion, vascular tumor embolus); other rare histologies which are treated as per the guidelines of this protocol may be allowed with approval of the medical monitor
* Concurrent monochemotherapy with cisplatin
* Radiation therapy to 70 Gray (Gy) to gross tumor in 2 Gy per fraction over 7 weeks using intensity modulated radiation therapy (IMRT) techniques for patients with intact tumors, and 60 Gy - 66 Gy in 2 Gy per fraction using IMRT for post-operative patients
* Induction chemotherapy (with up to 3 cycles of docetaxel and cisplatin based regimens) is allowed
* Ability to swallow and retain oral medication
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit normal (ULN)
* Calculated creatinine clearance >= 60 mL/min (Cockcroft-Gault equation)
* Patients of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Contraindication to full course chemoradiotherapy
* ECOG performance status >= 3
* Presence of distant metastatic disease
* Surgery with significant defect or flap in the oral cavity
* Poor dentition, ill-fitting dental appliances, obturators or any kind of resection prosthesis (can be enrolled if this can be corrected by a dentist prior to start of radiation therapy)
* Presence of other medical conditions causing mucositis (e.g., rheumatologic, severe gastroesophageal reflux, etc. at the discretion of the physician)
* Previous radiotherapy on head and neck district involving mucosa of oral cavity and/or oropharynx
* Use of chronic immunosuppressive drugs
* Brachytherapy or interstitial implantation treatment
* Other medical conditions that could make the patient not able to comply with the treatment
* Requirement of chronic steroid therapy (except when given for laryngeal edema)
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with severe mucositis (WHO score 3 or 4) | Up to 3 months after completion of study treatment
  The 2 treatment groups will be compared using the Mantel-Haenszel test, stratified by disease site and type of therapy, using a two-sided test at the alpha= 0.10 level of significance. Since emphasis is placed on the accurate estimation of treatment effect for use in the planning of a future confirmatory trial, corresponding estimates of effect size will also be computed along with 90% confidence intervals.

SECONDARY OUTCOMES:
Severity and duration of mucositis as assessed by dichotomized WHO Mucositis Global Severity Score (0-2 vs 3-4) and/or OMDQ scores | Up to 3 months after completion of study treatment
  The 2 treatment groups will be compared. The Mantel-Haenszel test, stratified by disease site and type of therapy, will be used for these comparisons.
Quality of life as assessed by EORTC QLQ-C30 questionnaire (with 1 being not at all and 4 being very much) | Up to 3 months after completion of study treatment
  The 2 treatment groups will be compared. Will be analyzed using Mann-Whitney U tests. All secondary analyses will be carried out using two-sided tests at the 10% level of significance.
Quality of Life as assessed by EORTC QLQ Head and Neck Cancer-Specific Module function and symptom sub-scores between groups (with 1 being not at all and 4 being very much) | Up to 3 months after completion of study treatment
  The 2 treatment groups will be compared. Will be analyzed using Mann-Whitney U tests. All secondary analyses will be carried out using two-sided tests at the 10% level of significance.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, Principal Investigator — Roswell Park Cancer Institute